CLINICAL TRIAL: NCT03459898
Title: Assessment of Left-sided Cardiac Sparing Through the Use of 3-dimensional Surface Matching-based Deep Inspiration Breath Hold and Active Breathing Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Irene Karam, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 268-2017
Record Dates: First submitted 2018-02-02; First posted 2018-03-09 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Left-Sided Breast Cancer
MeSH Terms: conditions — Unilateral Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Breathing Control (Other): To review our institutional clinical experience of applying the AlignRT system to monitor patient setup and reproducibility when using ABC and DIBH techniques in the treatment of left-sided breast cancer patients.
  Interventions: Device: AlignRT system (VisionRT Ltd., London, UK)
- Deep Inspiration Breath Hold (Other): To review our institutional clinical experience of applying the AlignRT system to monitor patient setup and reproducibility when using ABC and DIBH techniques in the treatment of left-sided breast cancer patients.
  Interventions: Device: AlignRT system (VisionRT Ltd., London, UK)

INTERVENTIONS:
Device: AlignRT system (VisionRT Ltd., London, UK) — To review our institutional clinical experience of applying the AlignRT system to monitor patient setup and reproducibility when using ABC and DIBH techniques in the treatment of left-sided breast cancer patients.

SUMMARY:
The standard treatment for breast cancer is surgery followed by adjuvant breast radiation therapy in most cases. For left sided breast cancers, the heart dose delivered by the radiation treatment is often of particular concern. In order to spare the heart, different strategies are currently available, including active breathing control (ABC) and voluntary deep in inspiration breath hold (DIBH) (both strategies are currently being used at our centre). To perform accurate heart-sparing treatments, it is important to ensure that patients are positioned consistently. One available approach is through surface imaging which tracks the position of a portion of the skin surface, known as the AlignRT system (VisionRT Ltd, London, UK).

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of left-sided breast malignancy
* Women who require left chest wall or breast irradiation status post mastectomy or lumpectomy
* Treatment with modified wide tangents to include IMCs
* Treatment with four-field technique
* Age >18 years
* Performance status ECOG <3
* Patient must be able to maintain a 30 second breath hold
* Conventional chest wall or breast radiation delivery dose of 50Gy/25 or hypofractionated chest wall/breast radiation delivery dose of 42.56Gy/16 with or without a boost

Exclusion Criteria:

* Right sided breast cancer patients
* Treatment with partial breast irradiation
* Previous left breast/chest wall irradiation
* Locally advanced breast cancer
* Pregnant patients
* Unable to follow commands

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Reproducibility of ABC or vDIBH set-up as measured by Align RT. | 2 years
  Reproducibility of set-up will be evaluated by determining discrepancies in patient's surface between treatment and CT simulation which will be acquired with the Align RT system using multiple measures along with daily portal images during treatment and weekly CBCTs.
Mean heart dose as determined using Align RT. | 2 years
  Estimate the change in mean heart dose for each breath-hold/heart sparing strategy by:
  i. Converting differences in heart position on 2D portal images acquired during treatment to 3D volumes on Pinnacle plans.
  ii. Using the CBCT images (acquired weekly), to recalculate dose to heart based on the patient's position and anatomy that day.

SECONDARY OUTCOMES:
The impact of Align RT with vDIBH as compared to vDIBH without AlignRT on quality of life as assessed by the EORTC core QoL questionnaire. | 2 years
  QoL will be assessed using the EORTC core QoL questionnaire (QLQ-C30) which is a well-validated and widely used QoL questionnaire available in multiple languages (12,13). QLQ-C30 is composed of 30 questions that represent 5 functional scales (physical, role, cognitive, emotional and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), and a global health / QoL scale. The questionnaire will be completed by patients at time of radiation simulation as baseline, at completion of RT (during routine review) and at the 6-8 week follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No